CLINICAL TRIAL: NCT01178515
Title: Impact of Low Fat Milk Intake on Cardiovascular Risk Indicators in Children 6-13 Years of Age
Brief Title: Low Fat Milk Intake and Cardio Vascular Risk (CVR) Indicators in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Dr. Salvador Villalpando, Instituto Nacional de Salud Publica
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Milk, Cardiovas risk, children; 1-865-6540 (Other: Ethics Committee, Instituto Nacional Salud Pub, Mexico)
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Cardiovascular Diseases
Keywords: epidemiological risk; diet; fat intake
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full fat milk (Sham Comparator): Full fat milk contain 3% fat
  Interventions: Other: Modification of the content of fat in milk
- Partially defatted milk (Experimental): Partially defatted milk contains 2% of fat
  Interventions: Other: Modification of the content of cows milk
- Defatted milk (Experimental): Defatted milk contains 1% fat
  Interventions: Other: Modification of the fat content of cows´ milk

INTERVENTIONS:
Other: Modification of the content of fat in milk — Comparison of three levels of fat content in cow´s milk
  Other Names: Liconsa milk
  Arms: Full fat milk
Other: Modification of the content of cows milk — Comparison of three levels of fat content in cows' milk
  Other Names: Liconsa low fat milk
  Arms: Partially defatted milk
Other: Modification of the fat content of cows´ milk — Comparison of three levels of fat content in cow´milk
  Other Names: Liconsa defatted milk
  Arms: Defatted milk

SUMMARY:
Substituting whole milk intake for defatted milk will improve indicators of cardiovascular risk, i.e. total cholesterol, triglycerides, Low Density Lipoprotein (LDL) and High Density Lipoprotein (HDL)cholesterol, apolipoproteins: ApoB100, Lp(a) and ApoA in a sample of Mexican children 6-13 years of age.

DETAILED DESCRIPTION:
Double blind trial in 600 children 6-13 years of age residing in 12 boarding schools. Schools will be randomized to distribute three types of milk namely: full fat milk (3% fat), partially defatted milk (2% fat) or defatted milk (1% fat) for 90 days of effective exposure (4 months total duration). Subjects will receive 400 mL of the corresponding milk every day (200 mL breakfast and 200 mL night meal) from Monday through Friday. During week ends they will eat a freely chosen diet at home. Milk intake will be measured every day. Diet by 24 h-recall. will be evaluated every month. Blood samples will be obtained at the beginning and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Attending selected boarding schools

Exclusion Criteria:

* No lactose intolerance

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 650 (Actual)
Dates: Start 2010-09; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk indicators | 4 months
  Cardiovascular risk is indicated by several determinations of blood fats namely: Total cholesterol, triglicerides, Low-density lipoprotein (LDL) and High density lipoprotein (HDL) cholesterol, lipoproteins: Apo a1,Apo B100 and Lp(a)

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Villalpando, MD, Ph D, Principal Investigator — Instituto Nacional de Salud Publica, Mexico; Teresa Shamah, M. Sc., Study Chair — Instituto Nacional de Salud Publica, Mexico; Yaveth Lara, M Sc, Study Chair — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- Comisíon para el Desarrollo de Pueblos Indigenas, Pachuca, Hidalgo, Mexico

REFERENCES:
- [Background] Stevens G, Dias RH, Thomas KJ, Rivera JA, Carvalho N, Barquera S, Hill K, Ezzati M. Characterizing the epidemiological transition in Mexico: national and subnational burden of diseases, injuries, and risk factors. PLoS Med. 2008 Jun 17;5(6):e125. doi: 10.1371/journal.pmed.0050125. PMID 18563960
- [Background] Berenson GS, Srinivasan SR, Bao W, Newman WP 3rd, Tracy RE, Wattigney WA. Association between multiple cardiovascular risk factors and atherosclerosis in children and young adults. The Bogalusa Heart Study. N Engl J Med. 1998 Jun 4;338(23):1650-6. doi: 10.1056/NEJM199806043382302. PMID 9614255
- [Background] Freedman DS. Clustering of coronary heart disease risk factors among obese children. J Pediatr Endocrinol Metab. 2002 Sep-Oct;15(8):1099-108. doi: 10.1515/JPEM.2002.15.8.1099. PMID 12387507
- [Background] Aguilar-Salinas CA, Gomez-Perez FJ, Rull J, Villalpando S, Barquera S, Rojas R. Prevalence of dyslipidemias in the Mexican National Health and Nutrition Survey 2006. Salud Publica Mex. 2010;52 Suppl 1:S44-53. doi: 10.1590/s0036-36342010000700008. PMID 20585729
- [Background] Corvalan C, Uauy R, Kain J, Martorell R. Obesity indicators and cardiometabolic status in 4-y-old children. Am J Clin Nutr. 2010 Jan;91(1):166-74. doi: 10.3945/ajcn.2009.27547. Epub 2009 Nov 18. PMID 19923378
- [Background] Villalpando S, Carrión C, Barquera S, Olaiz G, Robledo R. The body mass index is associated with hyperglycemia and alterations of some components of the metabolic syndrome in Mexican adolescents aged 10-19 years. Salud Pub Mex 2007; 49:s324-s330.
- [Background] Webber LS, Srinivasan SR, Wattigney WA, Berenson GS. Tracking of serum lipids and lipoproteins from childhood to adulthood. The Bogalusa Heart Study. Am J Epidemiol. 1991 May 1;133(9):884-99. doi: 10.1093/oxfordjournals.aje.a115968. PMID 2028978